CLINICAL TRIAL: NCT00279929
Title: Assessing the Effects of Dehydroepiandrosterone Replacement on the Mood of Adrenalectomised/Hypoadrenal Subjects
Brief Title: DHEA Replacement in Adrenalectomized/Hypoadrenal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 669-02; P01AG014383 (NIH)
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Aging; Dehydroepiandosterone Replacement; DHEA Replacement

INTERVENTIONS:
Procedure: DHEA Replacement

SUMMARY:
The role of dehydroepiandosterone (DHEA) and its sulphated ester (DHEAS) [together known as DHEA(S)] in humans remains to be fully elucidated. They are the most abundant circulating steroid hormones in humans with the principle source of production being the adrenal glands. In adrenalectomised or hypoadrenal subjects it is not standard clinical practice to replace this hormone. Whilst this lack of DHEA(S) is clearly not life threatening, the published literature on the psychological effects of replacement in this population has shown some benefit in quality of life but data concerning the metabolic effects is conflicting and incomplete. We wish to carry out a study to measure the effect of DHEA(S) replacement in a group of adrenalectomised / hypoadrenal subjects and measure the outcome of a number of psychological and metabolic parameters both prior to and after twelve weeks of 50 mg/day DHEA(S) in a double blind randomised cross over design.

Mood, quality of life and sexual well being will be assessed using validated questionnaires. In addition, we will utilise the GCRC facility to measure body composition using total body water and DEXA. We will measure insulin sensitivity, exercise performance, muscle fatigability and VO2 max. Pre- and post- intervention muscle biopsies will assess DHEA(S) effects on myosin heavy chain isoform expression; skeletal muscle mitochondrial ATP production and be used to assess muscle enzyme levels.

ELIGIBILITY:
Inclusion criteria:

* Subjects who have been adrenalectomised or have been hypoadrenal (from whatever cause) for > 24 months;
* Subjects who have been on a steady glucocorticoid replacement regime for >12 months;
* Women of child bearing age in whom oestrogen status has been steady for > 6 months - i.e. either on or off the oral contraceptive pill for that time;
* Subjects on other forms of hormone replacement therapy (e.g. thyroxin) in whom dose has remained the same for > 6 months.

Exclusion criteria:

* BMI >35 Kg/m2;
* Individuals with fasting blood glucose above 120mg/dl;
* A history of sex hormone dependant malignancy;
* A history of liver disease;
* Renal failure;
* Cardiovascular disease (other than hypertension);
* Polycythaemia;
* Pregnancy or breastfeeding;
* Cerebrovascular disorders;
* Neurological disorders;
* PSA levels above the age related reference range;
* Use of drugs known to alter mood within the 6 months prior to enrolment;
* Any drug known to affect hepatic biotransformation;
* Evidence of psychiatric disease or dementia;
* Postmenopausal women who have been on hormone replacement therapy for less than six months.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2002-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
physical performance (VO2 peak, muscle strength as measured by chest press, double knee extension, and isokinetic knee extension
quality of life
glucose and insulin metabolism
muscle protein synthesis
body composition

CONTACTS AND LOCATIONS:
Overall Officials: K. Sreekumaran Nair, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Dhatariya KK, Greenlund LJ, Bigelow ML, Thapa P, Oberg AL, Ford GC, Schimke JM, Nair KS. Dehydroepiandrosterone replacement therapy in hypoadrenal women: protein anabolism and skeletal muscle function. Mayo Clin Proc. 2008 Nov;83(11):1218-25. doi: 10.4065/83.11.1218. PMID 18990320